CLINICAL TRIAL: NCT03342612
Title: Cerebral Microstructural and Functional Changes After Single and Repeated Mild Traumatic Brain Injury
Brief Title: Multimodal Neuroimaging Analysis After Mild Traumatic Brain Injury
Acronym: CHANGE-TBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in including Mild Traumatic Brain Injury (mTBI) group despite an extended inclusion period of an additional 12 months
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX2016/07
Record Dates: First submitted 2017-08-03; First posted 2017-11-17 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Magnetic resonance imaging (MRI) to assess cerebral blood flow using Arteria Spin Labelling (ASL), structural changes using Diffusion Tensor Imaging (DTI), susceptibility weighted imaging (SWI), and functional changes using BOLD resting-functional MRI.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brain Magnetic Resonance Imaging (MRI) (Experimental): Neuroimaging protocol to assess brain changes after minor head trauma and over the time.
  Interventions: Procedure: Brain Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Brain Magnetic Resonance Imaging (MRI)

SUMMARY:
Mild Traumatic Brain Injury (mTBI), including concussion, is a real public health problem. Indeed mTBI might induce long-term brain disorders with increased risk of neurodegenerative diseases and the healthcare costs can be significant for both the individual and the society. However mTBI is called the "silent epidemic", because of the lack of research in this field in France as well as in the rest of the world. Most of the time, mTBI is associated with sports injuries, road traffic accidents and falls. The risk of neurodegenerative diseases is significantly increased with the repetition of mTBI, which may have a cumulative effect. In this context, playing football (or 'soccer') is associated with a high risk of concussion and with frequent head-ball contacts which are repeated during the training and matches. Moreover, football is the most popular team sport in the world, with more than 265 million players. The long-term impact of "heading" in football is still debated in the literature. Nevertheless, several studies suggest the possible emergence of early neurocognitive disorders. Otherwise, while mTBI is usually characterized by normal brain images using traditional neuroimaging techniques, microscopic anatomical changes might be detectable by new neuroimaging techniques. According to recent studies, cognitive dysfunctions could be based on these microstructural changes in the gray matter and white matter, secondary to the primary mechanical injury. Studies that have examined the structural changes in the brain white matter in football players are rare and lack of evidence regarding the consequences of accumulated brain impacts explains the lack of preventive measures in this sport. In addition, post-traumatic secondary lesions cause functional alterations of the neurovascular unit and its effect on cerebral perfusion may play a crucial role, which has never been yet explored in humans over the long term.

In this research, the investigators will develop a unique multi-modal neuroimaging protocols to assess brain changes after minor head trauma and over the time. Investigators want to perform magnetic resonance imaging (MRI) to assess cerebral blood flow using Arteria Spin Labelling (ASL), structural changes using Diffusion Tensor Imaging (DTI), susceptibility weighted imaging (SWI), and functional changes using BOLD resting-functional MRI.

ELIGIBILITY:
Inclusion Criteria:

Applicable to all :

- Male 18 to 25 years, enrolled in French Social Security.

Group of mTBI patients:

- Diagnosis of mTBI in the last 2 weeks confirmed in emergency department of Bordeaux CHU, using the WHO definition (2004): "head trauma ≤ 24h with Glasgow Coma Scale score of 13-15 and with one or more of the three symptoms following: confusion or disorientation, loss of consciousness for 30 minutes or less, posttraumatic amnesia for less than 24h".

Group of footballers:

- Member of the "CFA" and "U19" teams of "Girondins de Bordeaux".

Group of controls:

- Practicing regular physical activity (excluding combat or contact sports).

Exclusion Criteria :

* Abnormal neurological examination
* Drug addiction including alcohol Taking drugs targeting the central nervous system History of head trauma, or other notion of central nervous system injury
* History of severe high blood pressure, diabetes, chronic cardiovascular pathology, progressive or debilitating disease
* Subject unable to give informed consent
* Contraindication to MRI: head circumference> 60 - Claustrophobia - Pacemaker, Implantable Neurostimulation, Implantable Defibrillator - Cochlear Implants - Ocular or cerebral ferromagnetic foreign body
* Refusal to be informed of an abnormality detected during MRI.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy (FA) measure | Month 0
  Fractional anisotropy (FA) measure by Magnetic Resonance Imaging
Fractional anisotropy (FA) measure by Magnetic Resonance Imaging | Month 12
  Fractional anisotropy (FA) measure by Magnetic Resonance Imaging
Radial diffusivity (RD) measure | Month 0
  Radial diffusivity (RD) measure by Magnetic Resonance Imaging
Radial diffusivity (RD) measure | Month 12
  Radial diffusivity (RD) measure by Magnetic Resonance Imaging
Mean diffusivity (MD) measure | Month 0
  Mean diffusivity (MD) measure by Magnetic Resonance Imaging
Mean diffusivity (MD) measure | Month 12
  Mean diffusivity (MD) measure by Magnetic Resonance Imaging
Axial diffusivity (AD) measure | Month 0
  Axial diffusivity (AD) measure by Magnetic Resonance Imaging
Axial diffusivity (AD) measure | Month 12
  Axial diffusivity (AD) measure by Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Brain areas on MRI sequences | Month 0
Brain areas on MRI sequences | Month 12
Brain's white matter injury volume on MRI | Month 0
Brain's white matter injury volume on MRI | Month 12
Micro-bleedings measure | Month 0
  Micro-bleedings measure on MRI in the brain parenchyma
Micro-bleedings measure | Month 12
  Micro-bleedings measure on MRI in the brain parenchyma
Blood brain circulation on MRI | Month 0
Blood brain circulation on MRI | Month 12
Connectivity modification of on MRI | Month 0
Connectivity modification of on MRI | Month 12
Actimetry | Month 0
Actimetry | Month 12
Cognitive performances and emotional state by Ecological Momentary Assessment (EMA) | Month 0
Cognitive performances and emotional state by Ecological Momentary Assessment (EMA) | Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No